CLINICAL TRIAL: NCT01277809
Title: Community Alliance for Quality of Life in Long Term Care: The Effects of a Walking Program on Balance, Falls and Well Being in Individuals Residing in Long-term Care
Brief Title: The Effects of a Walking Program on Balance, Falls and Well Being in Individuals Residing in Long-term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Lilian Thorpe, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIO-BEB 10-125
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Accidental Falls; Muscle Weakness; Gait, Unsteady; Depression; Behavior
Keywords: Long term care; Aging; Accidental Falls; Muscle Weakness; Gait; Physical Fitness; Muscle Strength; Postural Balance; Activities of Daily Living; Body Weight; Blood Pressure; Depression; Behavior; Dementia
MeSH Terms: conditions — Muscle Weakness; Gait Disorders, Neurologic; Depression; Behavior; Body Weight; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): Participants will receive care as usual (Usual Care Group; UCG) that is provided by their long-term care unit.
- Interpersonal Interaction (Active Comparator): Participants will receive stationary 1:1 interaction time with the same research personnel who conduct the third group walking session at each individual care facility in order to control for the interpersonal interaction likely to be involved in the walking program. This group will receive the equivalent interpersonal interaction time with research personnel as those participating in the walking group. This interaction time will occur with the participant stationary, rather than walking with the researcher.
  Interventions: Behavioral: Interpersonal Interaction
- Walking Program (Experimental): Participants will walk five times per week under the supervision of a licensed physiotherapist.
  Interventions: Behavioral: Walking Program

INTERVENTIONS:
Behavioral: Interpersonal Interaction — Participants will receive stationary 1:1 interaction time with the same research personnel who conduct the third group walking session at each individual care facility in order to control for the interpersonal interaction likely to be involved in the walking program (Interpersonal Interaction Group; IIG). This group will receive the equivalent interpersonal interaction time with research personnel as those participating in the WPG group. This interaction time will occur with the participant stationary, rather than walking with the researcher.
  Arms: Interpersonal Interaction
Behavioral: Walking Program — Participants will walk five times per week, supervised by a licensed physiotherapist. Subjects will in general gradually increase their daily supervised walking time as tolerated to a maximum of 30 minutes once per day. The distance and number of minutes walked each time will be recorded. Interpersonal interaction will occur during the walking sessions, and will be similar in quality and quantity to that during the Interpersonal Interaction Group.
  Arms: Walking Program

SUMMARY:
The purpose of this study is to assess the effectiveness of a regular walking program (which inevitably involves human interaction) compared to a usual care condition and to a human interaction condition (without the extra walking program) in individuals residing in Long-Term Care (LTC). Outcomes of interest include: balance, strength, mobility, endurance, walking distance; rate and severity of falls; activities of daily living; mood and behaviour.

It is hypothesized that participants taking part in the walking program will demonstrate maximal benefits compared to the no treatment control group (usual care) and the participants who will only receive social interaction. It is expected that benefits of the walking program will include decreased fall rates, and improved balance, endurance, strength, mood, behaviour, activities of daily living and quality of life indices. Given research findings that the addition of pleasant activities improves resident mood (Teri et al, 1997; 2003), it is expected that participants in the social interaction only group will demonstrate improvements in mood and other indices of quality of life.

DETAILED DESCRIPTION:
Residents in LTC facilities in the Saskatoon Health Region and Regina Qu'Appelle Region will be recruited.

Inclusion criteria: Male or female residents who are able to follow simple instructions, who can ambulate with or without a walking aid for at least 10 meters, and who are willing to participate in the study procedures will be eligible to participate in the study.

Exclusion criteria: Residents who have experienced a recent cardiovascular event (within past 6 months) or have severe arthritis, cardiac instability, a vestibular disorder, uncontrolled hypertension, uncontrolled epilepsy, a recent fracture (past 4 months), who have had a recent admission into an acute care facility (past 4 months), who are scheduled for surgery or hospitalization in next 6 months or who are participating in another regular exercise program (three or more times per week) aimed at improving balance or strength will be excluded from the study.

Based on the sample size calculations, a sample size of 129 participants will provide ample power for the repeated measures analyses. Data will be collected from an additional 50 participants in order to deal with the possibility of attrition. Thus, total sample size is 179 participants.

The investigators will meet with the LTC facilities' administrators and staff to inform them of the study, inclusion and exclusion criteria, study procedures and interventions. They will be provided with copies of a one page information form which includes a space for residents (or substitute medical decision-maker, if appropriate) to indicate their signed consent to be approached by research staff with more detailed information (Appendix). Staff will provide this form to potential/eligible subjects, and will collect these forms when completed. Subjects who have consented to be contacted by research staff will be provided with more detailed information about the study by the research coordinator. If the resident is in agreement, he or she will then give written consent and will be entered into the study. The consent will include written permission for researchers to consult with the subject's family physician about the subject's health, and to ensure optimization of vitamin D intake prior to enrollment.

Although some subjects may have cognitive problems, the majority of subjects will be clearly competent to provide their own consent. However, some subjects may have more advanced cognitive problems than others and may therefore not fully appreciate the consequences of participation. In this situation the person who normally provides consent for medical treatment will provide appropriate consent. When capacity to provide full, informed consent is not clear, both the subject and the substitute decision-maker will be asked to sign the consent forms.

6. Procedures:

Step 1: Baseline assessment. All participants regardless of group will undergo the following assessments. The assessment of the outcome measures will be conducted by trained study personnel who will be blinded to group allocation.

1. The Senior Fitness Test (SFT). The SFT, a six-item battery that includes measures of dynamic upper and lower extremity strength and flexibility, aerobic endurance, and dynamic balance and agility will be completed ).
2. The Berg Balance Scale (BBS). The BBS, a tool currently being used in the RRMC, is a 14-item battery intended to objectively assess a person's ability to safely perform several common daily living tasks.
3. Grip Strength. Grip strength of the dominant and non-dominant hand-held dynamometer will be measured. Strength will be tested 3 times with each hand and the maximum score will be recorded.
4. Gait speed (6 metre walk test). Participants will be asked to walk a distance of 6 metres over a portable, computerized walkway (the GAITRite® system. An additional two metres of walking will be added at the beginning and end of the walkway to accommodate for acceleration and deceleration. Subjects will be asked to walk along the walkway. Gait parameters, including gait speed, will be recorded.
5. OARS Physical Activities of Daily Living (PADL) Sub-Scale. The OARS-PADL is a brief, valid, and reliable instrument that is used as a clinical assessment of functional status. The OARS-PADL will be completed by the research assistant with information provided by subjects' care provider.
6. Cornell Scale for Depression in Dementia (CSDD). Mood will be assessed using the CSDD, a well- validated, scale (based on caregiver reports) designed for the assessment of depression in individuals with dementia and individuals residing in long-term care. The CSDD will be completed by the research assistant with information provided by subjects' care provider.
7. The Geriatric Depression Scale (GDS) short form will be also used to assess self-identified depressive symptoms during the study.
8. Revised Memory and Behavior Problems Checklist (RMBPC). Behavioral problems will be assessed with the use of the RMBPC, a 24-item report that measures observable behavioral and memory problems. The RMBPC will be completed by the research assistant with information provided by subjects' care provider.
9. Short Portable Mental Status Questionnaire (SPMSQ).
10. Coloured Analogue Pain Scale is being used to assess pain via patient self-report.
11. Height, weight and other body measurements. We will measure height, knee-floor height, weight and waist, upper arm and calf circumference.
12. Vital signs including blood pressure. We will measure lying and standing blood pressure as well as heart rate and respiratory rate.

The participant's family physician will be asked to optimize vitamin D level of participants at baseline according to Canadian guidelines, as this can impact fall risk. This will involve measuring the Vitamin D level at baseline, and ordering Vitamin D 1,000 units daily if the participant is not already taking this.

Step 2: Randomization into one of three groups:

1. Participants will receive care as usual (Usual Care Group; UCG) that is provided by their long-term care unit.
2. Participants will receive stationary 1:1 interaction time with the same research personnel who conduct the third group walking session at each individual care facility in order to control for the interpersonal interaction likely to be involved in the walking program (Interpersonal Interaction Group; IIG). This group will receive the equivalent interpersonal interaction time with research personnel as those participating in the WPG group. This interaction time will occur with the participant stationary, rather than walking with the researcher.
3. Participants will participate in the Walking Program Group (WPG), in which a daily supervised walking program will be provided by study personnel. After randomization to the walking group, a licensed physiotherapist will first review test results and overall functioning, then develop a safe plan for a therapeutic walking program. This plan will include a protocol for termination and resumption of walking in case of physical symptoms such as shortness of breath, lightheadedness or chest pain. In situations of unexpected medical symptoms, the supervising staff nurse of the nursing unit will be consulted, who may suggest termination of the walking, or interim modification of the walking plan until reviewed by medical and physiotherapy staff. Subjects will in general gradually increase their daily supervised walking time as tolerated to a maximum of 30 minutes once per day, Monday to Friday. The distance and number of minutes walked each time will be recorded. Interpersonal interaction will occur during the walking sessions, and will be similar in quality and quantity to that during the Interpersonal Interaction Group.

Participants will wear a gait belt during all and with walking (if in the walking program group) and will be closely monitored by the research assistant who will be trained in safety issues.

Step 3: Subjects will participate in a four month intervention, as outlined in Step 2 above.

Step 4: After 2 months of the intervention (outlined in Step 2 above), all subjects will be re-tested as per baseline assessment (Step 1) with the exception of height and knee-floor height.

Step 5: After 4 months of intervention (outlined in Step 2 above), all subjects will be re-tested as per baseline assessment (Step 1) with the exception of height and knee-floor height.

Step 6: At 2 months and 4 months post-intervention, all subjects will be re-tested as per baseline assessment (Step 1) with the exception of height and knee-floor height.

A. In order to control for confounding variables and to characterize the sample, the following data will be extracted from the chart, including the chart copy of admission, date of admission, personal health number and most recent quarterly Minimum Data Set (MDS), by research personnel. The MDS is a computerized long-term care assessment system designed to improve the care given to long-term care residents, and has been utilized province-wide since 2001. Personal identifying information will only be extracted for the purpose of accurate linking to other study information, and will be removed prior to data analysis.

Data to be collected: date of birth, race/ethnicity, gender, highest level of education, diagnoses on admittance, medications, health conditions (CHESS Scale: health instability); Cognitive Performance Scale; Depression Rating Scale; Index of Social Engagement; ADL Self-Performance Hierarchy Scale; Pain; Continence; Oral/Nutritional status; Communication; Mood and Behaviour Patterns; Physical Functioning and Structural problems; Activity Pursuit Patterns; Special Treatments and Procedures.

B. Record of Falls: The incidence and nature of falls will be prospectively collected from the standard Saskatoon Health Region falls documentation for the period of the intervention (4 months) and for 4 months following intervention. Copies of falls documentation will be made from the clinical chart every week by study personnel.

Any participants' health concerns (identified by the participant and/or nursing staff) will be reviewed by the research coordinator and discussed with the Medical Safety Committee as appropriate.

7. Time Period (indicate the dates when the research project is expected to begin and to be completed. A final status report must be filed with the Ethics Office once data collection from the last subject is complete. The Ethics Office should be notified once the study site is closed.):

Anticipated start date is December 2010. We anticipate the study will take about 2 years to complete. Expected completion date is December 31, 2016.

8. Data Storage (In accordance with recommended guidelines provide a statement outlining the procedures you will use to store securely the research data. State how long and where the data will be stored and identify the person who will be assuming responsibility for data storage):

Study participant information will be stored according to HIPA guidelines. All documents and data collection forms will be stored in the School of Physical Therapy, in a locked filing cabinet in the office of Vanina Dal Bello-Haas (P.I.) for the required 10-year period. Signed consent forms will be stored separately from the study data in locked files. Study subjects will be identified by research study number only. Only study numbers and aggregate information will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults residing in a long term care facility
* Able to follow simple instructions
* Can ambulate with or without a walking aid for at least 10 meters
* Willing to participate in the study procedures Exclusion Criteria:

Exclusion criteria:

* Cardiovascular event within past 6 months
* Severe arthritis
* Clinical significant vestibular disorder
* Uncontrolled hypertension
* Uncontrolled epilepsy
* Fracture within the past 4 months
* Admission into an acute care facility in last 4 months
* Scheduled for surgery or hospitalization in next 6 months
* Already participating in another regular exercise program (three or more times per week) aimed at improving balance or strength

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2010-12; Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Falls | Eight months
  The incidence and nature of falls will be prospectively collected using a simple daily Fall Diary for the period of the intervention (4 months) and for 4 months following intervention. The Fall Diary will be kept at the residents' bedside and will staff will be asked to record the nature and location of the fall, activity and symptoms at the time of the fall, type of footwear, injuries resulting from the fall. Diaries will be collected every week by study personnel.

SECONDARY OUTCOMES:
Fitness | Eight months
  The Senior Fitness Test (SFT) (Rikli & Jones 1999a; 1999b) will assess dynamic upper and lower extremity strength and flexibility, aerobic endurance, and dynamic balance and agility.
Balance | Eight months
  The Berg Balance Scale will be used to objectively assess a person's ability to safely perform several common daily living tasks
Grip Strength | Eight months
  Grip strength of the dominant and non-dominant hand-held dynamometer will be measured. Strength will be tested 3 times with each hand and the maximum score will be recorded
Gait speed | Eight months
  Participants will be asked to walk a distance of 6 metres over a portable, computerized walkway (the GAITRite® system (CIR Systems Inc., Clifton, NJ). An additional two metres of walking will be added at the beginning and end of the walkway to accommodate for acceleration and deceleration. Subjects will be asked to walk along the walkway. Gait parameters, including gait speed, will be recorded.
Physical Activities of Daily Living | Eight months
  OARS Physical Activities of Daily Living (PADL) Sub-Scale (Fillenbaum 1988)will be used as a clinical assessment of functional status. The OARS-PADL will be completed by the research assistant with information provided by subjects' care provider.
Depression | Eight months
  Mood will be assessed using the Cornell Scale for Depression in Dementia, a well- validated scale designed for the assessment of depression in individuals with dementia and individuals residing in long-term care. The CSDD will be completed by the research assistant with information provided by subjects' care provider.
Behavioral problems | Eight months
  Behavioral problems will be assessed with the use of the Revised Memory and Behavior Problems Checklist (RMBPC), a 24-item report that measures observable behavioral and memory problems (Appendix). The RMBPC will be completed by the research assistant with information provided by subjects' care provider.
Vital signs | Eight months
  We will measure lying and standing blood pressure as well as heart rate and respiratory rate at baseline and every two months throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian U Thorpe, MD, PhD, Principal Investigator — University of Saskatchewan; Vanina Dal Bello-Haas, Ph. D, P.T., Principal Investigator — McMaster University
Locations (1):
- Saskatoon Health Region, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Kalu ME, Dal Bello-Haas V, Hadjistavropoulos T, Thorpe L, Griffin M, Ploeg J, Richardson J. The Effects of a Walking Intervention on Gait Parameters in Older Adults Residing in Long-Term Care: A Randomized Controlled Trial. J Nutr Health Aging. 2021;25(9):1099-1105. doi: 10.1007/s12603-021-1683-6. PMID 34725668
- [Derived] Dal Bello-Haas VP, Thorpe LU, Lix LM, Scudds R, Hadjistavropoulos T. The effects of a long-term care walking program on balance, falls and well-being. BMC Geriatr. 2012 Dec 18;12:76. doi: 10.1186/1471-2318-12-76. PMID 23249431